CLINICAL TRIAL: NCT05978973
Title: Elemental Diet and Gut Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Bianca Chang, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00002455:
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Food, Formulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- elemental diet (Experimental): subjects will be using the elemental diet packets daily. Subjects who are positive for excessive methane (i.e. methane level>10 ppm) will be required to complete a single daily fasting methane measurement (SMM) for the duration of the 14 days.
  Interventions: Dietary Supplement: Elemental Diet

INTERVENTIONS:
Dietary Supplement: Elemental Diet — . Elemental diets contain all daily required vitamins, micronutrients and macronutrients. The ingredients are readily digestible (carbohydrates, amino acids and medium chain fatty acids) and are absorbed within the proximal small bowel. One main disadvantage of elemental diets such as Vivonex is their unpalatability3 which has limited their use.

SUMMARY:
he primary objective of this study is to assess changes in stool microbiome profiles in patients after an elemental diet.

DETAILED DESCRIPTION:
The gut microbiome is the collection of microbes residing inside the gastrointestinal (GI) tract. The involvement of the gut microbiome has been demonstrated in multiple diseases processes including irritable bowel syndrome, small intestinal bacterial overgrowth (SIBO), Crohn's disease, and ulcerative colitis among many other diseases. A "healthy" diverse gut microbiome is associated with a better response to infections and immunopathogenic insults.

Many factors can affect the gut microbiome including medications, age, disease states and diet. Among these factors, diet is the easiest factor that can be modified to improve the gut microbiome. However, conducting dietary trials is challenging due to the inability to fully standardize what subjects eat even with strict dietary instructions. Moreover, individual preferences/allergies, the source of dietary ingredients, freshness, and food preparation are important steps which affect the diet and are challenging to standardize among subjects in a diet trial. This has led to significant ambiguity regarding the true extent and depth of dietary modifications on gut microbiome.

Apart from vitamins and micronutrients, the three main food macronutrients in the human diet are carbohydrates, protein and fat. Upon digestion, carbohydrates are broken into monosaccharides, proteins into amino acids and fats mainly into fatty acids. Elemental diets contain all daily required vitamins, micronutrients and macronutrients. The ingredients are readily digestible (carbohydrates, amino acids and medium chain fatty acids) and are absorbed within the proximal small bowel. One main disadvantage of elemental diets such as Vivonex is their unpalatability which has limited their use. A palatable elemental diet can be a very valuable tool to enable us to assess the effects of diet on the gut microbiome as it bypasses several confounding effects in dietary trials such as food allergies, individual digestion variability, completeness of the diet ingredients, and food preparation.

SIBO is a condition in which the gut microbiome plays an integral role and is defined by abnormal and excessive numbers of bacteria in the small bowel.4 Interest in SIBO has been fueled by the ever-increasing awareness of the human microbiome and its potential relationships to human health and disease. SIBO is a preferred condition to assess the effects of elemental diet on the gut microbiome, given the known role of the gut microbiome in SIBO. Those with SIBO experience a range of intestinal and extraintestinal symptoms including diarrhea, nausea, bloating, abdominal pain, and excess gas.

Commonly, SIBO has been defined by two methods: direct culture of small bowel aspirates, and indirect assessment using carbohydrate (e.g. lactulose or glucose) breath testing. SIBO is generally treated with antibiotics. Low fermentable and elemental diets also have positive effects in SIBO. Based on the potential effects of diet on the gut microbiome, we hypothesize that a two-week period of an elemental diet can change the gut microbiome in SIBO subjects.

ELIGIBILITY:
Inclusion Criteria:

* • Participant must be able to understand and provide informed consent

  * Males and Females ≥18-85
  * Female subjects of childbearing potential must have a negative pregnancy test upon study entry
  * Female (and male) subjects with reproductive potential, must agree to use FDA approved methods of birth control for the duration of the study
  * Subject self-reports experiencing SIBO symptoms within 30 days
  * Positive (abnormal) lactulose breath test for SIBO on visit 1 (day -7) as defined as:

    * Rise of hydrogen ≥ 20ppm within 90 minutes on LBT OR
    * A methane level ≥10 ppm at any point during the 120-minute LBT

Exclusion Criteria:

* • Inability or unwillingness of a participant to give written informed consent or comply with study protocol

  * Pregnancy or lactating
  * Type 1 or type 2 diabetes
  * Active or ongoing infection that requires antibiotics other than the participants known prophylactic medications (i.e. active infection or antibiotic use in the last 1 month)
  * Any condition that, in the opinion of the investigator, contraindicates participation in this study will be excluded from study participation.
  * History of known Phenylketonuria (PKU) disease
  * Non-English-speaking participants

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-06 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
assess changes in stool microbiome profiles | 28 DAYS
  is to assess changes in stool microbiome profiles in patients after an elemental diet, as determined by 16S rRNA gene sequencing • Microbiome profiles will be determined in stool samples provided on visit 2 (day 0), visit 4 (day 14) and visit 6 (day 28). These analyses will be performed in batch at the end of the study and the profiles at visit 4 (day 14) and visit 6 (day 28) will be compared to those at visit 2 (day 0).

CONTACTS AND LOCATIONS:
Overall Officials: Bianca Chang, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pimentel M, Mathur R, Wang J, Chang C, Hosseini A, Fiorentino A, Rashid M, Pichetshote N, Basseri B, Treyzon L, Chang B, Leite G, Morales W, Weitsman S, Kraus A, Rezaie A. A Smartphone Application Using Artificial Intelligence Is Superior To Subject Self-Reporting When Assessing Stool Form. Am J Gastroenterol. 2022 Jul 1;117(7):1118-1124. doi: 10.14309/ajg.0000000000001723. Epub 2022 Mar 14. PMID 35288511
- [Background] Wu X, Zhu Y, Yang M, Zhang J, Lin D. Biological responses of Eisenia fetida towards the exposure and metabolism of tris (2-butoxyethyl) phosphate. Sci Total Environ. 2022 Mar 10;811:152285. doi: 10.1016/j.scitotenv.2021.152285. Epub 2021 Dec 18. PMID 34933047
- [Background] Moore DA, Schatz D. Overprecision increases subsequent surprise. PLoS One. 2020 Jul 8;15(7):e0227084. doi: 10.1371/journal.pone.0227084. eCollection 2020. PMID 32639957
- [Background] Kilic E, Tennstedt P, Hogner A, Lebok P, Sauter G, Bokemeyer C, Izbicki JR, Wilczak W. The zinc-finger transcription factor SALL4 is frequently expressed in human cancers: association with clinical outcome in squamous cell carcinoma but not in adenocarcinoma of the esophagus. Virchows Arch. 2016 Apr;468(4):483-92. doi: 10.1007/s00428-016-1908-y. Epub 2016 Jan 27. PMID 26818834
- [Background] Rubin R. Botulinum Toxin to Treat Endometriosis Pain. JAMA. 2019 Aug 27;322(8):716. doi: 10.1001/jama.2019.12350. No abstract available. PMID 31454029
- [Background] Rotovnik Kozjek N, Kompan L, Zagar T, Mrevlje Z. Influence of enteral glutamine on inflammatory and hormonal response in patients with rectal cancer during preoperative radiochemotherapy. Eur J Clin Nutr. 2017 May;71(5):671-673. doi: 10.1038/ejcn.2017.11. Epub 2017 Mar 8. PMID 28272402
- [Background] Pimentel M, Constantino T, Kong Y, Bajwa M, Rezaei A, Park S. A 14-day elemental diet is highly effective in normalizing the lactulose breath test. Dig Dis Sci. 2004 Jan;49(1):73-7. doi: 10.1023/b:ddas.0000011605.43979.e1. PMID 14992438
- [Background] Gombert A, Van Herzeele I. We Want to OPERATE! Eur J Vasc Endovasc Surg. 2020 May;59(5):775. doi: 10.1016/j.ejvs.2020.01.033. Epub 2020 Feb 20. No abstract available. PMID 32088068
- [Background] Speller B, Metcalfe K, Kennedy ED, Facey M, Greenblatt E, Scheer AS, Warner E, Joy AA, Wright FC, Baxter NN. The "Begin Exploring Fertility Options, Risks and Expectations" (BEFORE) decision aid: development and alpha testing of a fertility tool for premenopausal breast cancer patients. BMC Med Inform Decis Mak. 2019 Oct 28;19(1):203. doi: 10.1186/s12911-019-0912-y. PMID 31660965
- [Derived] Rezaie A, Chang BW, de Freitas Germano J, Leite G, Mathur R, Houser K, Hosseini A, Brimberry D, Rashid M, Mehravar S, Villanueva-Millan MJ, Sanchez M, Weitsman S, Fajardo CM, Rivera IG, Joo L, Chan Y, Barlow GM, Pimentel M. Effect, Tolerability, and Safety of Exclusive Palatable Elemental Diet in Patients With Intestinal Microbial Overgrowth. Clin Gastroenterol Hepatol. 2025 Nov;23(12):2306-2317.e7. doi: 10.1016/j.cgh.2025.03.002. Epub 2025 Apr 4. PMID 40189034